CLINICAL TRIAL: NCT04238559
Title: Use of the SWAMECO Questionnaire in the General Population to Detect Swallowing Difficulties
Brief Title: Use of the SWAMECO Questionnaire Basel
Acronym: SWAMECO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02187
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Swallowing Difficulties
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self-report questionnaire — Fill in the SWAMECO questionnaire

SUMMARY:
A patient self-report questionnaire was developed that assesses subjective swallowing difficulties with medication intake, the SWAMECO questionnaire. It was validated in a highly specific population and will now be tested in the general population.

DETAILED DESCRIPTION:
Based on a systematic literature review, a novel self-report questionnaire was developed in 2016 to assess subjective swallowing difficulties with medication intake and their practical consequences in ambulatory patients, the SWAMECO questionnaire. It consists of 30 items divided into 5 sections Complaints, Intensity, Localization, Coping strategies, and Adherence to medication. It was validated in people suffering from systemic sclerosis (SSc), a rare multisystem autoimmune disease that often leads to swallowing problems with food and liquids with progression. The aim of this study is now to validate the questionnaire in the general population. Patients presenting in the community pharmacy with a prescription of at least 3 different medications for a minimum of 3 months will fill in the questionnaire on site.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more
* is living in the community setting
* is receiving three or more medications for a period not less than three months, independently of the frequency of the intake

Exclusion Criteria:

* patients who are not able to provide written conformed consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project population is the general population.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
swallowing difficulties assessed by Questionnaire | 5 minutes
  The variable of primary interest is the answer to the question number 4: "Do you experience swallowing difficulties when you take your medicines?"

SECONDARY OUTCOMES:
medication adherence assessed by Questionnaire | 5 minutes
  Answers to q 26-28: "how many days did you miss at least one dose of any of your medicines?", "how good a job did you do at taking your medicines in the way you were supposed to?", "how often did you take your medicines in the way you were supposed to?"

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnet, Dr., Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No